CLINICAL TRIAL: NCT04901065
Title: Xylocaine to Freeze During Unpleasant Nasopharyngeal Swabs: a Randomized, Double-Blinded, Placebo Controlled-Trial
Brief Title: Xylocaine to Freeze During Unpleasant Nasopharyngeal Swabs
Acronym: Xylofuns
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Evelyne D.Trottier (Other)
Responsible Party: Sponsor-Investigator, Evelyne D.Trottier, MD, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-3414
Record Dates: First submitted 2021-05-14; First posted 2021-05-25 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research assistant enrolling the patients was blinded to treatment assignment because he did not know to which bottle the patient was randomized (A or B) and he did not know what was contained in the bottle
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xylocaine (Experimental): The study intervention was the administration of 10 mg of intranasal lidocaine in one nostril using 1 spray of 0.1mL of a 10% lidocaine solution 5 minutes before NPS. This was done using the standard long nozzle.
  Interventions: Drug: Xylocaine
- Control (Sham Comparator): The control group received the placebo with the same application technique using an empty bottle of lidocaine 10% with the same long nozzle for delivery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xylocaine — The study intervention was the administration of 10 mg of intranasal lidocaine in one nostril using 1 spray of 0.1mL of a 10% lidocaine solution 5 minutes before NPS. This was done using the standard long nozzle
  Other Names: Xylocaine spray
  Arms: Xylocaine
Drug: Placebo — The control group received the placebo with the same application technique using an empty bottle of lidocaine 10% with the same long nozzle for delivery
  Arms: Control

SUMMARY:
Since the beginning of the COVID-19 pandemic, nasopharyngeal swabs (NPS) have been recommended to detect the virus. This procedure has been reported to be painful by 85% of children The aim of the study was to assess whether pretreatment with topical lidocaine reduces the discomfort experienced by children during a nasopharyngeal swab.

This was a RCT among children aged 8-17 years old who need a NPS. The primary outcome was pain intensity as measured by the Visual Analog Scale .

ELIGIBILITY:
Inclusion:

* 6-17 years old inclusively
* Children for whom a NPS was ordered

Exclusion:

* Children presenting with the following acute conditions, which could either prevent the lidocaine from being properly administered, or pose a risk for the patient as increased absorption of the medication might occur:

  * Nasal or airway burns, trauma or major anomaly
  * Cardiorespiratory compromise
* Children for whom an informed consent could not be obtained

  * Any other life-threatening condition or priority one patient requiring emergency support
  * Language barrier
* Children presenting with conditions that could prevent their ability to reliably report their pain:

  * Severe intellectual disability
  * Severe pain upon presentation
  * Administration of opiates prior to the NPS
* Children presenting with the following chronic conditions, which could either prevent the lidocaine from being properly administered, or pose a risk for the patient:

  * Hypersensitivity/allergy to the medication or a known component
  * Methemoglobinemia
  * G6PD deficiency
  * Familial malignant hyperthermia
  * Pseudocholinesterase deficiency
  * Severe hepatic impairment
  * Severe cardiac condition or use of antiarrhythmic medication
  * Risk of airway aspiration

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Pain during the procedure | During procedure
  Self-reported pain immediately after the NPS as measured using a validated self-reported pain scale: the Visual Analog Scale (VAS

SECONDARY OUTCOMES:
Anxiety during the procedure | During procedure
  ● Evaluation of fear prior to the administration of the study intervention and the NPS using the Children's Fear Scale
Discomfort | During procedure
  Discomfort at administration of the study intervention using a yes/no question
Pain 2 NRS | During procedure
  Evaluation of pain immediately after the NPS using a clinically relevant tool, the verbal Numeric Rating Scale
Number of patients with physical restriction | During procedure
  Evaluation of the patient position (sitting, lying down, standing) and if physical restraints was done (none, redirection of movements, comfort position/minimal comfortable restriction or actively restrain) to perform the swab and to which extent
Utility according to nurses | During procedure
  ● Triage nurses evaluation on the efficiency of the intervention in reducing pain in the patient, using a likert scale of 1 to 5
Adverse event | 48 hours following intervention
  Adverse effects reported by caregivers in the 24-48hrs following administration of medication
Desire to reuse the intervention in a futur procedure, at follow up | 48 hours following intervention
  Asking caregivers in the 24-48hrs following intervention if they would recommend the intervention before a NPS as standard of care for pediatric patients. Yes/no question.

CONTACTS AND LOCATIONS:
Locations (1):
- Evelyne D Trottier, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No